CLINICAL TRIAL: NCT02016352
Title: Cerebrospinal Fluid Proteome in Hydrocephalus
Acronym: PROLIPHYC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10 045 08; 2011-A01091-40 (Other: AFSSAPS ID-RCB)
Record Dates: First submitted 2013-06-18; First posted 2013-12-20 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2020-11

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: hydrocephalus; proteomic; cerebrospinal fluid
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient (Experimental): patient CSF extraction with hydrocephalus
  Interventions: Biological: patient CSF extraction with hydrocephalus
- witness (Other): patient without hydrocephalus but with peridural catheter for anesthetic. Witness CSF extraction has realized on catheter.
  Interventions: Biological: witness CSF extraction

INTERVENTIONS:
Biological: patient CSF extraction with hydrocephalus — CSF extraction
  Arms: patient
Biological: witness CSF extraction — CSF extraction from patient not suffering from hydrocephalus
  Arms: witness

SUMMARY:
PROLIPHYC is a collaborative prospective study that aims at discovering deep cerebrospinal fluid (CSF) proteome with a new clinically-compatible proteomics strategy, in a cohort of 100 patients suspected of neurodegenerative diseases and/or normal pressure hydrocephalus.

DETAILED DESCRIPTION:
CSF proteome is the real time protein content that may reveal useful biomarkers for diagnosis and therapeutic decision-making. But the low protein concentration in CSF and the low volumes typically obtained after lumbar puncture precludes the conventional use of proteomic analysis. We miniaturized the method to be compatible with low-volume samples by combination of nanoLC-MS/MS analysis and combinatorial peptide ligand library technology to reduce the dynamic range of protein concentration in CSF and unmask previously undetected proteins. We demonstrated that this deep proteomic analysis allows profiling the CSF proteome with a reasonable depth, in short analytical times and good accuracy. We settled a clinically-compatible proteomics strategy targeting the deep CSF proteome discovery.

The PROLIPHYC study is a prospective study that aims at analysing CSF proteome with our new strategy in a cohort of patients suspected of normal pressure hydrocephalus and/or related neurodegenerative diseases. The PROLIPHYC project combines detailed clinical and neuropsychological evaluation, gait analysis, MRI brain imaging, lumbar CSF dynamics and deep proteome. We hypothesize in the PROLIPHYC study that a specific cluster of polypeptides can be associated with Alzheimer disease, vascular dementia and normal pressure hydrocephalus profiles. Validating this hypothesis might be a significant step towards a proteomic lexicon of aging brain, neurodegenerative diseases and dementia.

Neurosciences department and Alzheimer disease centre from the Toulouse University Hospital are both involved in this project. The deep proteomic study is performed in Toulouse by the Institute of Pharmacology and Structural Biology with the academic support of the Institute of Mathematics of Toulouse.

ELIGIBILITY:
Inclusion Criteria:

* Gait problems, cognitive decline, urinary incontinence and enlarged ventricles on imaging

Exclusion Criteria:

* Psychiatric disorders
* Lumbar punction contraindication
* RMI contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
CSF proteome measure | 48 hours
  CSF extraction (3 ml)

SECONDARY OUTCOMES:
correlation between CSF proteome and gait analysis | 72 hours
  compare results from CSF proteome and gait analysis
correlation between CSF proteome and MRI brain imaging | 72 hours
  compare results from CSF proteome and brain imaging

CONTACTS AND LOCATIONS:
Overall Officials: Eric SCHMIDT, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Guillotin S, Vallet A, Lorthois S, Cestac P, Schmidt E, Delcourt N. Association Between Homocysteine, Frailty and Biomechanical Response of the CNS in NPH-Suspected Patients. J Gerontol A Biol Sci Med Sci. 2022 Jul 5;77(7):1335-1343. doi: 10.1093/gerona/glac074. PMID 35325129
- [Result] Vallet A, Del Campo N, Hoogendijk EO, Lokossou A, Baledent O, Czosnyka Z, Balardy L, Payoux P, Swider P, Lorthois S, Schmidt E. Biomechanical response of the CNS is associated with frailty in NPH-suspected patients. J Neurol. 2020 May;267(5):1389-1400. doi: 10.1007/s00415-019-09689-z. Epub 2020 Jan 29. PMID 31997040
- [Result] Guillotin S, Fulzele A, Vallet A, de Peredo AG, Mouton-Barbosa E, Cestac P, Andrieu S, Burlet-Schiltz O, Delcourt N, Schmidt E. Cerebrospinal fluid proteomic profile of frailty: Results from the PROLIPHYC cohort. Aging Cell. 2024 Jul;23(7):e14168. doi: 10.1111/acel.14168. Epub 2024 May 2. PMID 38698559